CLINICAL TRIAL: NCT04077190
Title: Extension Study of Protocol RC-001b- Safety and Efficacy of Adult Adipose-Derived Stem Cell Injection Into Partial Thickness Rotator Cuff Tears
Brief Title: Safety and Efficacy of Adult Adipose-Derived Stem Cell Injection Into Partial Thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC-003
Record Dates: First submitted 2019-08-23; First posted 2019-09-04 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- adipose-derived stem cell injection (Experimental): Ultrasound guided injection of 5cc adipose derived stem cells
  Interventions: Device: Adipose-derived stem cells
- cortisone injection (Active Comparator): Ultrasound guided injection of cortisone
  Interventions: Device: cortisone injection

INTERVENTIONS:
Device: Adipose-derived stem cells — 5cc adipose derived stem cells.
  Arms: adipose-derived stem cell injection
Device: cortisone injection — cortisone injection
  Arms: cortisone injection

SUMMARY:
Extension Study of Protocol RC-001- Safety and Efficacy of Adult Adipose-Derived Stem Cell Injection into Partial Thickness Rotator Cuff Tears. Purpose is to investigate the Long- term safety and efficacy of autologous stem cells in patients with partial thickness rotator cuff tears versus a steroid treatment.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate the safety and superior effectiveness in functional improvement in patients with partial-thickness rotator cuff tears (PTRCTs) after the administration of a single injection of adipose-derived regenerative cells (ADRCs) into the partial-thickness rotator cuff tear compared to the administration of a single corticosteroid injection into the associated subacromial space.

The ADRC mixture is generated from the Transpose® RT System, a point-of-care solution for extraction of an autologous regenerative cell mixture from the adipose tissue after a same-day limited liposuction procedure. A pilot clinical study was recently completed using an injection of ADRC compared to a corticosteroid injection for treatment of PTRCTs. Results support the initiation of a pivotal study to study the same.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed participation in RC-001 (NCT02918136) study
* Must have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures associated with this trial.

Exclusion Criteria:

* none

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Long term Safety as indicated through adverse event rate between ADSC and TAU arms | at 24 months
  Adverse event rate
Long term Safety as indicated through adverse event rate between ADSC and TAU arms | at 36 months
  Adverse event rate
Long term efficacy of pain and function through Short Form-36 Shoulder Score health questionnaires | at 24 months
  Short form-36 score compared to baseline (total score = 800)
Long term efficacy of pain and function through Short Form-36 Shoulder Score health questionnaires | at 36 months
  Short form-36 score compared to baseline (total score = 800)
Long term efficacy of pain and function through ASES Shoulder Score health questionnaires | at 24 months
  ASES score compared to baseline (total score = 100)
Long term efficacy of pain and function through ASES Shoulder Score health questionnaires | at 36 months
  ASES score compared to baseline (total score = 100)

SECONDARY OUTCOMES:
Long term efficacy will be evaluated through MRIs pre- and post-injection for the therapeutic intent to treat a rotator cuff injury: Percentage improvement in tendon tear size and thickness | at 36 months
  Percentage improvement in tendon tear size and thickness

CONTACTS AND LOCATIONS:
Overall Officials: jason Hurd, MD, Principal Investigator — Sanford Orthopedics & Sports Medicine
Locations (2):
- United States (2):
  - Sanford Orthopedics and Sports Medicine - Fargo, Fargo, North Dakota
  - Sanford orthopedics and Sports Medicine - Sioux Falls, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No